CLINICAL TRIAL: NCT03018600
Title: Glucose Profiles of High-Dose Glucocorticoid Treatment in Young Patients With Diverse Autoimmune Disease With or Without Long-Term Low-Dose Glucocorticoid
Brief Title: Continuous Glucose Monitoring on Patients With Active Autoimmune Diseases Following High-dose Predisone Treatment
Acronym: CGM
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUMCH-ZS965
Record Dates: First submitted 2017-01-07; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-04

CONDITIONS: Glucocorticoid-induced Hyperglycemia
Keywords: prednisone, autoimmune disease
MeSH Terms: conditions — Autoimmune Diseases | interventions — Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The participants tested the patients' blood sample for insulin, C peptide, HbA1c, GA and other basic biochemical values (liver and renal function, lipid levels).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: We included 15 inpatients admitted to the Immunology Department, Peking Union Medical College Hospital (PUMCH), Beijing, China from April 1, 2016 to September 1, 2016.Intervention including glucocorticoid: 1-2mg/kg/day prednisone-equivalent (intravenous/oral methylpredisolone or oral prednisone) to the patients every morning at 8am for at least five days.
  Interventions: Behavioral: diet and exercise intervention
- 2: We included 10 inpatients admitted to the Immunology Department, Peking Union Medical College Hospital (PUMCH), Beijing, China from April 1, 2016 to September 1, 2016.Intervention including glucocorticoid: using less than 15mg/day prednisone-equivalent glucocorticoid maintenance for at least 3 months and now treating with 1-2mg/kg/day prednisone-equivalent (intravenous/oral methylpredisolone or oral prednisone) for the relapse of primary autoimmune disease for at least five days.
  Interventions: Behavioral: diet and exercise intervention

INTERVENTIONS:
Behavioral: diet and exercise intervention — consult nutrious doctors giving specific food and take regular exercise when under steroid therapy

SUMMARY:
Glucocorticoid is widely used in clinical treatment. Recently, there was research about glucose fluctuations under low-dose and pulse steroid therapy in elderly patients with active autoimmune diseases. Through this prospective trial, the investigators wanted to know the blood glucose characteristics under high dosage glucocorticoid (1-2 mg/kg/day prednisone or equivalent) in young patients (30-40 years) with active autoimmune diseases with or without low-dose glucocorticoid maintenance. The investigators used continuous glucose monitoring for 72 hours to get a better understanding of the glucose levels.

DETAILED DESCRIPTION:
As known to all, the dosage and duration of glucocorticoid influences the glucose levels in different diseases. Continuous glucose monitoring becomes a newly effective technology to better understand the glucose level. In this study,the investigators enrolled 25 patients with certain active autoimmune diseases during high-dosage glucocorticoid therapy at Peking Union Medical College Hospital. It was done by monitoring three-day continuous glucose levels by holding continuous glucose monitoring system underneath the skin, which helped to show a unique picture of fluctuations. The participants were divided into two groups according to the glucocorticoid therapy. Group 1 enrolled subjects who were newly commenced 1-2mg/kg/day prednisone-equivalent (intravenous/oral methylpredisolone or oral prednisone) for at least five days. Group 2 enrolled subjects who had underwent less than 15mg/day prednisone-equivalent glucocorticoid maintenance for at least 3 months but treated with high-dose glucocorticoid for the relapse during the study This finding is useful for the suitable treatment to control the hyperglycemia in young patients.

ELIGIBILITY:
Inclusion Criteria:

* Young patients with exacerbation of autoimmune disease, requiring 1-2mg/kg/day prednisone or equivalent for treatment;
* could undergo <15mg/kg/day prednisone or equivalent glucocorticoid maintenance in the previous three months;

Exclusion Criteria:

* patients with history of diabetes;
* patients with severe organ dysfunction or failure;
* patients with febrile conditions;

Ages: 25 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The subjects were recruited from inpatients admitted to the Immunology Department, Peking Union Medical College Hospital (PUMCH), Beijing, China from April 1, 2016 to September 1, 2016. Patients' primary disease was diagnosed according to the criteria by American College of Rheumatology. The spectrum of autoimmune disease included Systemic lupus Erythematosus (SLE), Connective tissue disorders, Sjogren Syndrome, Systemic sclerosis, IgG4-related disease, Bahcet's disease, ANCA-associated vasculitis, polymyositis, dermatomyositis.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
glucose values of 24 hours (mmol/L); | 72 hours CGMS monitoring

SECONDARY OUTCOMES:
the amounts of patients developing hyperglycemia | 72 hours CGMS monitoring

IPD SHARING:
Plan to Share IPD: No